CLINICAL TRIAL: NCT01631006
Title: Acute Hemodynamic Effects of Continous Positive Airway Pressure (CPAP) in Patients With Hypertrophic Cardiomyopathy
Brief Title: Effects of Continous Positive Airway Pressure (CPAP) in Hypertrophic Cardiomyopathy
Acronym: CPAPandHCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Geraldo Lorenzi-Filho, Associated Professor of Pulmonary Division, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SDC 325209/003
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Non-obstructive Hypertrophic Cardiomyopathy; Obstructive Hypertrophic Cardiomyopathy
Keywords: CPAP; Hypertrophic cardiomyopathy; Blood Pressure; The focus of the present study is to evaluate the acute hemodynamic effects of CPAP in patients with non-obstructive and obstructive hypertrophic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low CPAP pressure (Sham Comparator): Patients are submmited to a CPAP with low pressure for 20 minutes
  Interventions: Device: CPAP
- High CPAP pressure (Active Comparator): Patients are submmited to a high pressure of CPAP for 20 minutes
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — A low or high CPAP pressure is delivered for 20 minutes

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is the most common genetic cardiac disease, is a cause of disability including heart failure, atrial fibrillation, and sudden death, with an annual mortality varying from 1% to 6%. Obstructive sleep apnea (OSA) is extremely common among patients with established cardiovascular disease, including hypertension and atrial fibrillation and when present may contribute to worse cardiovascular outcome. Although patients with HCM do not necessarily have typical characteristics of patients with OSA, such as obesity and increasing age, there is recent evidence that OSA is extremely common among patients with HCM, with a prevalence ranging from 32% to 71%. The presence of OSA among patients with HCM is independently associated with worse structural and functional impairment of the heart, including atrial and aorta enlargement, worse New York Heart Association functional class, and worse quality of life. Therefore, the recognition and treatment of OSA is a new area of research that may impact in the management of patients with HCM.

ELIGIBILITY:
Inclusion Criteria:

* both genders
* over 18 years-old
* hemodynamically stable
* with no other cardiac disease
* consent form signed

Exclusion Criteria:

* presence of pacemaker
* spontaneous withdrawal
* previous cardiorespiratory arrest
* atrial fibrilation during echocardiography

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Cadiac performance by echocardiography | acutely

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Nerbass FB, Salemi VMC, Pedrosa RP, Portilho NP, Ferreira-Filho JCA, Moriya HT, Antunes MO, Arteaga-Fernandez E, Drager LF, Lorenzi-Filho G. Acute Effects of Nasal CPAP in Patients With Hypertrophic Cardiomyopathy. Chest. 2016 Nov;150(5):1050-1058. doi: 10.1016/j.chest.2016.05.004. Epub 2016 May 7. PMID 27167210